CLINICAL TRIAL: NCT04060615
Title: Properties of Myocardial Microcirculation in Patients With Different Pathomorphological Substrates, Before and After Recanalization of Coronary Artery Chronic Total Occlusion
Brief Title: Properties of Myocardial Microcirculation in Patients With Different Pathomorphological Substrates, Before and After Recanalization of Coronary Artery CTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Belgrade (Other)
Collaborators: Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Milan Dobric, Assistant professor, University of Belgrade
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 61206-1296/2-17
Record Dates: First submitted 2019-08-04; First posted 2019-08-19 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Chronic Total Occlusion of Coronary Artery
Keywords: chronic total occlusion; coronary flow reserve
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: All patients with chronic total occlusion will undergo the PCI procedure of the occlusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic total occlusion of the coronary artery (Other): In each patient before the PCI procedure, the investigators will assess myocardial viability, functional parameters of collateral blood vessels, and quality of life. 24h and 6 months after the procedure these parameters will be reevaluated as well as functional parameters of the treated coronary artery.
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — PCI of the chronic total occlusion of the coronary artery

SUMMARY:
This study will evaluate the changes in myocardial microcirculatory parameters of the collateral donor artery after recanalization of coronary artery chronic total occlusion.

DETAILED DESCRIPTION:
This study will include patients with chronic total occlusion (CTO) of one coronary artery who will undergo the recanalization of the CTO. Before the procedure, myocardial viability, ischemia, functional parameters of the collateral donor blood vessels, echocardiography, and quality of life will be assessed. After the recanalization, these parameters will be assessed again 24h and 6 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with signed informed consent to participate in the study
* Presence of one CTO on native coronary arteries (with TIMI 0 flow)
* Presence of clinical indication for attempting a PCI for CTO (at least one of the criteria present):

  1. Symptoms of typical stable angina
  2. Presence of inducible ischemia in the territory of the occluded artery
  3. Presence of viable myocardium in the territory of the occluded artery
* The diameter of the occluded artery ≥2.5mm

Exclusion Criteria:

* Acute coronary syndrome in the past month
* Existing contraindication for administration of dual antiplatelet therapy in the duration of 12 months
* Contraindications for implanting the drug-eluting stents
* Existence of 2 or more CTOs on native coronary arteries (with TIMI 0 flow)
* Severe tortuosity or calcifications of the coronary arteries
* Left ventricle aneurysm
* Previous coronary artery bay-pass graft or any other cardiac surgery
* Previous myocardial infarction in the coronary artery territory different from the CTO
* Ejection fraction of the left ventricle less than 30%
* Permanent atrial fibrillation
* Pregnancy
* Patients with known allergy to iodine contrast that cannot be controlled with medication
* Patients who are unable or unwilling to cooperate and come for check-up visits
* Life expectancy less than a year
* Hemorrhagic diathesis, coagulopathy, or rejection of blood transfusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-12-15 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Coronary flow reserve | six months
  Change in coronary flow reserve of the collateral donor vessel (after PCI as compared to values before PCI) will be regarded as primary outcome measure

SECONDARY OUTCOMES:
Coronary flow velocity reserve | six months
  Correlation of coronary flow velocity reserve change of the collateral donor vessel (after PCI as compared to values before PCI) with viability measured by the percentage of viable myocardium on Single Photon Emission Computed Tomography (SPECT) of myocardial perfusion.
Wall Motion Score Index (WMSI) | six months
  Relation of coronary flow velocity reserve change with wall motion score index on stres-echocardyography test where the wall motion segment abnormalities will be graded as such: 1 - normokinesis, 2 - hypokinesis, 3- akinesis and 4 dyskinesis, and the higher values indicates worse outcome
Change from Baseline Stable Angina questionnaire (SAQ) at 6 months | six months
  Relation of coronary flow velocity reserve change with the quality of life measured by 19-item Seattle Angina Questionnaire that assesses angina frequency (with 9 questions where answers range from 1 to 6, the total score ranges from 0 to 100, where the higher value indicates better outcome), angina stability ( with 1 question where answers range from 1 to 6, the total score ranges from 0 to 100, where the higher value indicates better outcome), the angina frequency scale (with 2 questions where answers range from 1 to 5, the total score ranges from 0 to 100, where the higher value indicates better outcome), treatment satisfaction (with 4 questions where answers range from 1 to 6, the total score ranges from 0 to 100, where the higher value indicates better outcome), and disease perception/QoL (with 3 questions where answers range from 1 to 5, the total score ranges from 0 to 100, where the higher value indicates better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Branko D Beleslin, MD, PhD, Study Director — University of Belgrade; Miodrag C Ostojic, MD, PhD, Study Director — University of Belgrade
Locations (1):
- Clinical Centre of Serbia, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sianos G, Werner GS, Galassi AR, Papafaklis MI, Escaned J, Hildick-Smith D, Christiansen EH, Gershlick A, Carlino M, Karlas A, Konstantinidis NV, Tomasello SD, Di Mario C, Reifart N; EuroCTO Club. Recanalisation of chronic total coronary occlusions: 2012 consensus document from the EuroCTO club. EuroIntervention. 2012 May 15;8(1):139-45. doi: 10.4244/EIJV8I1A21. No abstract available. PMID 22580257
- [Background] Delacretaz E, Meier B. Therapeutic strategy with total coronary artery occlusions. Am J Cardiol. 1997 Jan 15;79(2):185-7. doi: 10.1016/s0002-9149(96)00710-2. PMID 9193021
- [Background] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Background] Werner GS, Gitt AK, Zeymer U, Juenger C, Towae F, Wienbergen H, Senges J. Chronic total coronary occlusions in patients with stable angina pectoris: impact on therapy and outcome in present day clinical practice. Clin Res Cardiol. 2009 Jul;98(7):435-41. doi: 10.1007/s00392-009-0013-5. Epub 2009 Mar 18. PMID 19294443
- [Background] Fefer P, Knudtson ML, Cheema AN, Galbraith PD, Osherov AB, Yalonetsky S, Gannot S, Samuel M, Weisbrod M, Bierstone D, Sparkes JD, Wright GA, Strauss BH. Current perspectives on coronary chronic total occlusions: the Canadian Multicenter Chronic Total Occlusions Registry. J Am Coll Cardiol. 2012 Mar 13;59(11):991-7. doi: 10.1016/j.jacc.2011.12.007. PMID 22402070
- [Background] Rathore S, Matsuo H, Terashima M, Kinoshita Y, Kimura M, Tsuchikane E, Nasu K, Ehara M, Asakura Y, Katoh O, Suzuki T. Procedural and in-hospital outcomes after percutaneous coronary intervention for chronic total occlusions of coronary arteries 2002 to 2008: impact of novel guidewire techniques. JACC Cardiovasc Interv. 2009 Jun;2(6):489-97. doi: 10.1016/j.jcin.2009.04.008. PMID 19539251
- [Background] Saito S. Progress in angioplasty for chronic total occlusions again. Catheter Cardiovasc Interv. 2010 Nov 15;76(6):850-1. doi: 10.1002/ccd.22847. No abstract available. PMID 21104774
- [Background] Godino C, Sharp AS, Carlino M, Colombo A. Crossing CTOs-the tips, tricks, and specialist kit that can mean the difference between success and failure. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1019-46. doi: 10.1002/ccd.22161. PMID 19950136
- [Background] Werner GS. The role of coronary collaterals in chronic total occlusions. Curr Cardiol Rev. 2014 Feb;10(1):57-64. doi: 10.2174/1573403x10666140311123814. PMID 24611646
- [Background] Werner GS, Bahrmann P, Mutschke O, Emig U, Betge S, Ferrari M, Figulla HR. Determinants of target vessel failure in chronic total coronary occlusions after stent implantation. The influence of collateral function and coronary hemodynamics. J Am Coll Cardiol. 2003 Jul 16;42(2):219-25. doi: 10.1016/s0735-1097(03)00624-7. PMID 12875755
- [Background] Werner GS, Surber R, Kuethe F, Emig U, Schwarz G, Bahrmann P, Figulla HR. Collaterals and the recovery of left ventricular function after recanalization of a chronic total coronary occlusion. Am Heart J. 2005 Jan;149(1):129-37. doi: 10.1016/j.ahj.2004.04.042. PMID 15660044
- [Background] Werner GS, Surber R, Ferrari M, Fritzenwanger M, Figulla HR. The functional reserve of collaterals supplying long-term chronic total coronary occlusions in patients without prior myocardial infarction. Eur Heart J. 2006 Oct;27(20):2406-12. doi: 10.1093/eurheartj/ehl270. Epub 2006 Sep 26. PMID 17003048
- [Background] Werner GS, Fritzenwanger M, Prochnau D, Schwarz G, Ferrari M, Aarnoudse W, Pijls NH, Figulla HR. Determinants of coronary steal in chronic total coronary occlusions donor artery, collateral, and microvascular resistance. J Am Coll Cardiol. 2006 Jul 4;48(1):51-8. doi: 10.1016/j.jacc.2005.11.093. Epub 2006 Jun 12. PMID 16814648
- [Background] Werner GS, Ferrari M, Heinke S, Kuethe F, Surber R, Richartz BM, Figulla HR. Angiographic assessment of collateral connections in comparison with invasively determined collateral function in chronic coronary occlusions. Circulation. 2003 Apr 22;107(15):1972-7. doi: 10.1161/01.CIR.0000061953.72662.3A. Epub 2003 Mar 24. PMID 12665484
- [Background] Werner GS, Richartz BM, Gastmann O, Ferrari M, Figulla HR. Immediate changes of collateral function after successful recanalization of chronic total coronary occlusions. Circulation. 2000 Dec 12;102(24):2959-65. doi: 10.1161/01.cir.102.24.2959. PMID 11113046
- [Background] Werner GS, Emig U, Bahrmann P, Ferrari M, Figulla HR. Recovery of impaired microvascular function in collateral dependent myocardium after recanalisation of a chronic total coronary occlusion. Heart. 2004 Nov;90(11):1303-9. doi: 10.1136/hrt.2003.024620. PMID 15486127
- [Background] Zimarino M, Ausiello A, Contegiacomo G, Riccardi I, Renda G, Di Iorio C, De Caterina R. Rapid decline of collateral circulation increases susceptibility to myocardial ischemia: the trade-off of successful percutaneous recanalization of chronic total occlusions. J Am Coll Cardiol. 2006 Jul 4;48(1):59-65. doi: 10.1016/j.jacc.2005.12.079. Epub 2006 Jun 12. PMID 16814649
- [Background] Sachdeva R, Uretsky BF. The effect of CTO recanalization on FFR of the donor artery. Catheter Cardiovasc Interv. 2011 Feb 15;77(3):367-9. doi: 10.1002/ccd.22806. PMID 20853349
- [Background] Kurisu S, Mitsuba N, Ishibashi K, Kato Y, Dohi Y, Nishioka K, Kihara Y. A pitfall of fractional flow reserve associated with the presence of collateral circulation. Intern Med. 2011;50(22):2811-3. doi: 10.2169/internalmedicine.50.6104. Epub 2011 Nov 15. PMID 22082894
- [Background] Ladwiniec A, Hoye A. The haemodynamic effects of collateral donation to a chronic total occlusion: Implications for patient management. Int J Cardiol. 2015 Nov 1;198:159-66. doi: 10.1016/j.ijcard.2015.06.174. Epub 2015 Jul 6. PMID 26163908
- [Background] Ladwiniec A, Cunnington MS, Rossington J, Mather AN, Alahmar A, Oliver RM, Nijjer SS, Davies JE, Thackray S, Alamgir F, Hoye A. Collateral donor artery physiology and the influence of a chronic total occlusion on fractional flow reserve. Circ Cardiovasc Interv. 2015 Apr;8(4):e002219. doi: 10.1161/CIRCINTERVENTIONS.114.002219. PMID 25805570
- [Background] Spertus JA, Winder JA, Dewhurst TA, Deyo RA, Prodzinski J, McDonell M, Fihn SD. Development and evaluation of the Seattle Angina Questionnaire: a new functional status measure for coronary artery disease. J Am Coll Cardiol. 1995 Feb;25(2):333-41. doi: 10.1016/0735-1097(94)00397-9. PMID 7829785
- [Background] Pavlovic SV, Sobic-Saranovic DP, Beleslin BD, Ostojic MC, Nedeljkovic MA, Giga VL, Petrasinovic ZR, Artiko VM, Todorovic-Tirnanic MV, Obradovic VB. One-year follow-up of myocardial perfusion and function evaluated by gated SPECT MIBI in patients with earlier myocardial infarction and chronic total occlusion. Nucl Med Commun. 2009 Jan;30(1):68-75. doi: 10.1097/mnm.0b013e32831a40dd. PMID 19306516
- [Background] Gunning MG, Anagnostopoulos C, Davies G, Knight CJ, Pennell DJ, Fox KM, Pepper J, Underwood SR. Simultaneous assessment of myocardial viability and function for the detection of hibernating myocardium using ECG-gated 99Tcm-tetrofosmin emission tomography: a comparison with 201Tl emission tomography combined with cine magnetic resonance imaging. Nucl Med Commun. 1999 Mar;20(3):209-14. doi: 10.1097/00006231-199903000-00002. PMID 10093069
- [Background] Germano G, Kiat H, Kavanagh PB, Moriel M, Mazzanti M, Su HT, Van Train KF, Berman DS. Automatic quantification of ejection fraction from gated myocardial perfusion SPECT. J Nucl Med. 1995 Nov;36(11):2138-47. PMID 7472611
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Giga V, Dobric M, Beleslin B, Sobic-Saranovic D, Tesic M, Djordjevic-Dikic A, Stepanovic J, Nedeljkovic I, Artiko V, Obradovic V, Seferovic PM, Ostojic M. Estimation of infarct size using transthoracic Doppler echocardiographic measurement of coronary flow reserve in infarct related and reference coronary artery. Int J Cardiol. 2013 Sep 20;168(1):169-75. doi: 10.1016/j.ijcard.2012.09.099. Epub 2012 Oct 8. PMID 23058345
- [Background] Djordjevic-Dikic A, Beleslin B, Stepanovic J, Giga V, Tesic M, Dobric M, Stojkovic S, Nedeljkovic M, Vukcevic V, Dikic N, Petrasinovic Z, Nedeljkovic I, Tomasevic M, Vujisic-Tesic B, Ostojic M. Prediction of myocardial functional recovery by noninvasive evaluation of Basal and hyperemic coronary flow in patients with previous myocardial infarction. J Am Soc Echocardiogr. 2011 May;24(5):573-81. doi: 10.1016/j.echo.2011.01.004. PMID 21514503
- [Background] Beleslin B, Ostojic M, Djordjevic-Dikic A, Vukcevic V, Stojkovic S, Nedeljkovic M, Stankovic G, Orlic D, Milic N, Stepanovic J, Giga V, Saponjski J. The value of fractional and coronary flow reserve in predicting myocardial recovery in patients with previous myocardial infarction. Eur Heart J. 2008 Nov;29(21):2617-24. doi: 10.1093/eurheartj/ehn418. Epub 2008 Sep 30. PMID 18826987
- [Background] Baykan AO, Kalkan GY, Sahin DY, Elbasan Z, Gur M, Seker T, Turkoglu C, Cayli M. Coronary flow velocity reserve in donor artery and myocardial performance index after successful recanalization of chronic total coronary occlusions. J Invasive Cardiol. 2015 Jun;27(6):E75-81. PMID 26028662
- [Background] Schaper W. Collateral circulation: past and present. Basic Res Cardiol. 2009 Jan;104(1):5-21. doi: 10.1007/s00395-008-0760-x. Epub 2008 Dec 20. PMID 19101749
- [Background] Matsuo H, Kawase Y. Physiological impact of CTO recanalization assessed by coronary pressure measurement: a case report. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):E459-64. doi: 10.1002/ccd.24842. Epub 2013 Apr 11. PMID 23359324
- [Background] Iqbal MB, Shah N, Khan M, Wallis W. Reduction in myocardial perfusion territory and its effect on the physiological severity of a coronary stenosis. Circ Cardiovasc Interv. 2010 Feb 1;3(1):89-90. doi: 10.1161/CIRCINTERVENTIONS.109.904193. No abstract available. PMID 20160187
- [Background] Melikian N, Cuisset T, Hamilos M, De Bruyne B. Fractional flow reserve--the influence of the collateral circulation. Int J Cardiol. 2009 Mar 6;132(3):e109-10. doi: 10.1016/j.ijcard.2007.08.034. Epub 2007 Dec 4. PMID 18055036
- [Background] Sachdeva R, Agrawal M, Flynn SE, Werner GS, Uretsky BF. Reversal of ischemia of donor artery myocardium after recanalization of a chronic total occlusion. Catheter Cardiovasc Interv. 2013 Oct 1;82(4):E453-8. doi: 10.1002/ccd.25031. Epub 2013 Jul 3. PMID 23703834
- [Background] Watanabe H, Saito N, Matsuo H, Kawase Y, Watanabe S, Bao B, Yamamoto E, Higami H, Nakatsuma K, Kimura T. In vitro assessment of physiological impact of recipient artery intervention on the contralateral donor artery. Cardiovasc Revasc Med. 2015 Mar;16(2):90-100. doi: 10.1016/j.carrev.2015.01.003. Epub 2015 Jan 30. PMID 25870153
- [Background] Rentrop KP, Cohen M, Blanke H, Phillips RA. Changes in collateral channel filling immediately after controlled coronary artery occlusion by an angioplasty balloon in human subjects. J Am Coll Cardiol. 1985 Mar;5(3):587-92. doi: 10.1016/s0735-1097(85)80380-6. PMID 3156171
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784
- [Background] Hesse B, Lindhardt TB, Acampa W, Anagnostopoulos C, Ballinger J, Bax JJ, Edenbrandt L, Flotats A, Germano G, Stopar TG, Franken P, Kelion A, Kjaer A, Le Guludec D, Ljungberg M, Maenhout AF, Marcassa C, Marving J, McKiddie F, Schaefer WM, Stegger L, Underwood R. EANM/ESC guidelines for radionuclide imaging of cardiac function. Eur J Nucl Med Mol Imaging. 2008 Apr;35(4):851-85. doi: 10.1007/s00259-007-0694-9. PMID 18224320
- [Background] Wahba FF, Bavelaar-Croon CD, Baur LH, Zwinderman AH, van Roosmalen RP, Pauwels EK, van der Wall EE. Detection of residual wall motion after sustained myocardial infarction by gated 99Tcm-tetrofosmin SPECT: a comparison with echocardiography. Nucl Med Commun. 2001 Feb;22(2):175-82. doi: 10.1097/00006231-200102000-00009. PMID 11258404
- [Background] Acampa W, Cuocolo A, Petretta M, Bruno A, Castellani M, Finzi A, Gerundini P. Tetrofosmin imaging in the detection of myocardial viability in patients with previous myocardial infarction: comparison with sestamibi and Tl-201 scintigraphy. J Nucl Cardiol. 2002 Jan-Feb;9(1):33-40. doi: 10.1067/mnc.2002.118122. PMID 11845127
- [Derived] Dobric M, Beleslin B, Tesic M, Djordjevic Dikic A, Stojkovic S, Giga V, Tomasevic M, Jovanovic I, Petrovic O, Rakocevic J, Boskovic N, Sobic Saranovic D, Stankovic G, Vukcevic V, Orlic D, Simic D, Nedeljkovic MA, Aleksandric S, Juricic S, Ostojic M. Prompt and consistent improvement of coronary flow velocity reserve following successful recanalization of the coronary chronic total occlusion in patients with viable myocardium. Cardiovasc Ultrasound. 2020 Jul 21;18(1):29. doi: 10.1186/s12947-020-00211-4. PMID 32693812

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT04060615/Prot_SAP_000.pdf